CLINICAL TRIAL: NCT03632798
Title: Avastin Plus Chemotherapy vs. Avastin Plus Chemotherapy Chosen by Cancer Stem Cell Chemosensitivity Testing in the Management of Patients With Recurrent Platinum-Resistant or -Sensitive Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Cancer
Brief Title: Avastin Plus Chemotherapy vs. Avastin Plus Chemotherapy Guided by Cancer Stem Cell Test in Recurrent Ovarian Cancer
Acronym: ACSCO
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Cordgenics, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: CG02EOC
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Ovarian Cancer
Keywords: ChemoID; cancer stem cells; drug response assay; ovarian cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Intervention Model Description: parallel group randomized controlled clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Study investigators will be kept blind to the schedule. All participants will be screened by the ChemoID drug response assay; however, the treating physician will receive the ChemoID results only for those participants who are randomized to receive ChemoID-guided treatment arm.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physician Choice treatment (Active Comparator): Participants will be treated with control chemotherapy treatment (Bevacizumab plus standard-of-care chemotherapy chosen by the Physician from the provided list).
  Control chemotherapy treatment will be chosen from any of the following standard-of-care chemotherapy drugs or combinations:
  * Liposomal Doxorubicin;
  * Docetaxel;
  * Paclitaxel;
  * Carboplatin;
  * Cisplatin;
  * Gemcitabine;
  * Topotecan;
  * Carboplatin, Gemcitabine;
  * Cisplatin, Gemcitabine;
  * Carboplatin, Liposomal Doxorubicin;
  * Carboplatin, Paclitaxel;
  * Carboplatin, Docetaxel.
  The treating physician will NOT receive the ChemoID assay results from the ChemoID lab.
  Interventions: Diagnostic Test: ChemoID assay; Drug: Chemotherapy
- ChemoID-guided treatment (Experimental): Participants will be treated with Bevacizumab plus ChemoID-guided standard-of-care chemotherapy drugs from the provided list.
  ChemoID-guided treatment will be chosen from the following standard-of-care chemotherapy drugs or combinations:
  * Liposomal Doxorubicin;
  * Docetaxel;
  * Paclitaxel;
  * Carboplatin;
  * Cisplatin;
  * Gemcitabine;
  * Topotecan;
  * Carboplatin, Gemcitabine;
  * Cisplatin, Gemcitabine;
  * Carboplatin, Liposomal Doxorubicin;
  * Carboplatin, Paclitaxel;
  * Carboplatin, Docetaxel.
  The treating physician will receive the ChemoID assay results from the ChemoID lab.
  Interventions: Diagnostic Test: ChemoID assay; Drug: Chemotherapy

INTERVENTIONS:
Diagnostic Test: ChemoID assay — The ChemoID test is a CLIA-certified and CAP-accredited drug response assay performed by a hospital clinical pathology laboratory that uses patient's live tumor cells to indicate which chemotherapy agent (or combinations) will kill not only bulk of tumor cells, but importantly the cancer stem cells (CSCs) that are known to cause cancer to recur. During the assay, cancer stem cells and bulk tumor cells from an individual patient are exposed to FDA-approved chemotherapy drugs.
  The test measures the cytotoxic effect of actual doses of standard-of-care chemotherapies. The ChemoID drug response assay reports a prioritized list of effective and ineffective chemotherapies. The test is designed to target cancer stem cells to mitigate tumor relapse.
Drug: Chemotherapy — Chemotherapies chosen by Physician or ChemoID assay are in the same list of FDA approved drugs to treat recurrent ovarian cancer.
  Chemotherapy list:
  * Liposomal Doxorubicin;
  * Docetaxel;
  * Paclitaxel;
  * Carboplatin;
  * Cisplatin;
  * Gemcitabine;
  * Topotecan;
  * Carboplatin, Gemcitabine;
  * Cisplatin, Gemcitabine;
  * Carboplatin, Liposomal Doxorubicin;
  * Carboplatin, Paclitaxel;
  * Carboplatin, Docetaxel.
  Other Names: List of cytotoxic chemotherapy drugs

SUMMARY:
The purpose of this randomized clinical study is to confirm the utility of chemosensitivity (ChemoID) tumor testing on cancer stem cells as a predictor of clinical response in recurrent epithelial ovarian cancer (EOC), fallopian tube, or primary peritoneal cancer, regardless of platinum sensitivity.

Population studied will be female participants experiencing a 1st, 2nd, or 3rd recurrence of any stage epithelial ovarian cancer.

DETAILED DESCRIPTION:
This study is designed as a parallel group randomized controlled clinical trial to determine if recurrent Epithelial Ovarian Cancer (EOC) patients treated with Bevacizumab plus drugs predicted by the ChemoID assay will have better outcomes than patients treated with standard-of-care control therapy (Bevacizumab plus chemotherapy chosen by the Physician).

Upon obtaining informed consent, all eligible participants affected by 1st, 2nd, or 3rd relapse of EOC regardless of platinum sensitivity (both platinum sensitive and resistant) will have a tumor biopsy or a cancer-positive fluid collection sample to undergo ChemoID drug response testing with multiple FDA-approved chemotherapeutic agents.

Eligible participants will be randomized to a standard treatment arm with control treatment (Bevacizumab plus chemotherapy chosen by the Physician from the provided list), or to a study arm of Bevacizumab plus FDA-approved drugs selected by the ChemoID drug response assay.

A stratified randomization approach for treatment arm assignment will be used with strata based on relapse number, platinum sensitivity, and study site to ensure balance within these cells.

ELIGIBILITY:
Inclusion Criteria:

* 1. Informed consent obtained and signed;
* 2. Willing and able to commit to study procedures including long-term follow-up visit(s);
* 3. At least 18 years old at the time of enrollment;
* 4. Negative pregnancy test for women of childbearing potential
* 5. Experiencing 1st, 2nd, or 3rd recurrent epithelial ovarian cancer of any stage regardless of platinum sensitivity, (platinum-sensitive, -resistant, or -refractory);
* 6. Histopathological or cytological confirmation of recurrent epithelial ovarian carcinoma, peritoneal cancer or fallopian tube cancer.
* 7. Evaluable disease - defined as RECIST 1.1 measurable disease OR not measurable disease (defined as solid and/or cystic abnormalities on radiographic imaging that do not meet RECIST 1.1 definitions for target lesions OR ascites and/or pleural effusion that has been pathologically demonstrated to be disease-related in the setting of a CA125 > 2x ULN).
* 8. At least 30 days post-cytotoxic chemotherapy and/or monoclonal antibody therapy prior to enrollment;
* 9. Toxicities of prior therapy (excepting alopecia) should be resolved to less than or equal to Grade 1 as per CTCAE v4.0 (http://ctep.cancer.gov/protocol development/electronic_applications/ctc.htm). Patients with long-standing stable grade 2 neuropathy may be considered after discussion with the Study Chair.
* 10. ECOG Performance Status Score of ≤ 2, KPS≥70, or 0-1 GOG status
* 11. Adequate laboratory values within 60 days of enrollment to study defined as follows:

  1. WBC ≥ 3000/mm3
  2. Hgb ≥ 10 mg/dl
  3. Hct ≥ 28%
  4. Platelet count ≥ 100,000/μL
  5. Serum creatinine ≤ 2.0 mg/dl
  6. Total bilirubin ≤ 2.5 mg/dl
  7. AST/SGOT ≤ 3 times ULN. If intrahepatic liver metastases are present, AST and ALT must be ≤ 5 times institutional ULN.
  8. Random urine protein/creatinine ratio ≤ 1 or 24 hour urine protein < 0.1 gram.
* 12. Appropriate for tissue sampling either by tumor biopsy or peritoneal or pleural fluid collection.

Exclusion Criteria:

* 1. Estimated life expectancy of <6 months, as estimated by the investigator in consultation with participating oncologists;
* 2. Ovarian cancer of a low grade serous, mucinous, or clear cell histology;
* 3. Uncontrolled diabetes;
* 4. Patients with clinically significant proteinuria; urine protein should be screened by urine protein-creatinine ratio (UPCR); the UPCR has been found to correlate directly with the amount of protein excreted in a 24 hour urine collection; specifically, a UPCR of 1.0 is equivalent to 1.0 gram of protein in a 24-hour urine collection; obtain at least 4 ml of a random urine sample in a sterile container (does not have to be a 24-hour urine); send sample to lab with request for urine protein and creatinine levels (separate requests); the lab will measure protein concentration (mg/dL) and creatinine concentration (mg/dL); the UPCR is derived as follows: protein concentration (mg/dL)/creatinine (mg/dL); patients must have a UPCR ≤ 1.0 to allow participation in the study;
* 5. Symptomatic cardiac conditions;
* 6. Contraindications to bevacizumab including uncontrolled hypertension, known arterial or venous thromboembolism, known nephrotic syndrome, history of abdominal fistula, GIP, or intra-abdominal abscess; clinical signs or symptoms of GI obstruction and/or requirement for parenteral hydration or nutrition; nonhealing wound, ulcer, or bone fracture; bleeding diathesis or significant coagulopathy; known CNS disease, clinically significant cardiovascular disease; and a major surgical procedure within 28 days of enrollment or anticipated to occur while participating in study;
* 7. Enrollment in another clinical study that precludes allowing the oncologist to select chemotherapy regimens;
* 8. Previously participated in this study;
* 9. Any condition that would, in the opinion of the investigator, place the participant at an unacceptable risk, or render the participant unable to meet the requirements of the protocol (including long-term study follow-up).
* 10. Documented history of ovarian cancer of a low malignant potential phenotype or unclear cell histology.
* 11. CA-125 only disease without RECIST 1.1 measurable or otherwise evaluable disease
* 12. Patients may not use any complementary or alternative medicines including natural herbal products or folk remedies as they may interfere with the effectiveness of the study treatments.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Ovarian Cancer is a female disease
Enrollment: 0 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-06-10 (Actual); Study Completion 2019-06-10 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) | 36 months
  Progression free survival (PFS) in patients with recurrent epithelial ovarian cancer (EOC) who receive standard of care treatment (Bevacizumab plus chemotherapy chosen by the Physician from the provided list) versus Bevacizumab plus ChemoID drug response assay-directed chemotherapy.

SECONDARY OUTCOMES:
Median Overall Survival (OS) | 36 months
  Overall survival (OS) in patients with recurrent EOC who receive standard of care treatment (Bevacizumab plus chemotherapy chosen by the Physician from the provided list) versus Bevacizumab plus ChemoID drug response assay-directed chemotherapy.
Objective Tumor Response | 36 months
  ORR: partial or complete response by RECIST v1.1 (Response Evaluation Criteria In Solid Tumors)
HRQOL | 36 months
  Health-Related Quality of Life (HRQOL)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly J Wilkinson, MD, Principal Investigator — University of Mississippi Medical Center
Locations (3):
- United States (3):
  - Univeristy of Mississippi Medical Center, Jackson, Mississippi
  - Charleston Area Medical Center, Charleston, West Virginia
  - Edwards Comprehensive Cancer Center - Cabell Huntington Hospital, Huntington, West Virginia

IPD SHARING:
Plan to Share IPD: No